CLINICAL TRIAL: NCT07255287
Title: Behavioral Weight Loss Plus Sleep Health Program (BWL+SLEEP) Feasibility Pilot Study
Brief Title: Behavioral Weight Loss and Sleep Health Intervention
Acronym: DREAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-1317; 1K24HL169755 (NIH)
Record Dates: First submitted 2025-10-31; First posted 2025-12-01 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Overweight and Obese Adults
Keywords: overweight; obese; sleep; weight loss
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Weight Loss Program Plus Sleep Health Intervention (Experimental): Participants will receive a 6-month group-based behavioral weight loss intervention that incorporates strategies to improve sleep health.
  Interventions: Behavioral: BWL+Sleep

INTERVENTIONS:
Behavioral: BWL+Sleep — Participants will receive a 6-month group-based behavioral weight loss intervention that incorporates strategies to improve sleep health.

SUMMARY:
This is a 6-month single-arm pilot and feasibility study designed to examine if a behavioral weight loss (BWL) intervention with an added sleep health program (BWL+SLEEP) can achieve clinically meaningful weight loss and improvements in a composite sleep health score. The investigators will also evaluate the feasibility of recruitment and retention of study participants and will obtain feedback from participants to improve the program's incorporation of strategies to improve sleep health.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index 25-40 kg/m2
* Suboptimal sleep defined as: 1) short sleep duration (actigraphy total sleep time <6.5 hrs/night), 2) sleep irregularity (actigraphy standard deviation, SD of wake time, bed time or sleep duration >60 min), 3) poor sleep satisfaction/quality (Pittsburgh Sleep Quality Index, PSQI single item sleep quality question response of "fairly bad" or "very bad"), 4) suboptimal sleep timing (actigraphy sleep midpoint before 2 AM or after 4 AM), 5) daytime sleepiness (Epworth Sleepiness Scale, ESS >10) and/or 6) suboptimal sleep efficiency (actigraphy sleep efficiency <85%).
* Physically Inactive: defined as <150 minutes per week of exercise at moderate intensity or greater and <60 min per day of total habitual physical activity (i.e., work related, transportation related) at moderate intensity or greater, over the past 3 months.
* No self-report of acute or chronic disease (cardiovascular disease (CVD), diabetes, pulmonary, gastrointestinal disorders, and orthopedic problems in particular).
* No plans to relocate within the next 12 months.
* No plans for extended travel (>2 weeks) within the next 12 months.
* Live or work within 30 minutes of the AHWC (exceptions may be made at the discretion of the Study PI).
* Capable and willing to give informed consent, understand exclusion criteria, and accept the randomized group assignment.
* Own or willing to purchase a smartphone, willing to download and use the Oura Ring and/or Headspace App if randomized to these components. (Data from the Pew Research Center 2024 Mobile Fact Sheet suggests >95% of adults in our target age range own a smartphone)
* Have a primary care physician (or are willing to establish care prior to study enrollment) to address any medical issues which may arise during screening procedures or study interventions.
* No contraindications to exercise or limitations on ability to be physically active.
* Agree to refrain from use of anti-obesity medications (AOMs) agents during the 6-month pilot study.
* For Females:

  * Not currently pregnant or lactating,
  * Not pregnant within the past 6 months,
  * Not planning to become pregnant in the next 12 months. Sexually active women of childbearing potential may be enrolled if they have had a tubal ligation or use a reliable means of contraception.

Exclusion Criteria:

* Diastolic blood pressure >100 mmHG, systolic blood pressure >160 mmHG, or resting heart rate >100 bpm as measured in duplicate on the screening visit after 5 minutes of rest in a seated position.
* Diabetes (fasting glucose greater than or equal to 126 mg/dL or Hemoglobin A1C greater than or equal to 6.5%) as measured during the screening visit.
* Undiagnosed hypo- or hyper-thyroid (TSH outside of the normal range as measured during the screening visit) or history of uncontrolled thyroid disorder. History of thyroid disease or current thyroid disease treated with a stable medication regimen for at least 6 months is acceptable.
* Hematocrit, white blood cell count or platelets significantly outside the normal reference range as measured on the screening visit.
* Triglycerides >400 mg/dL as measured on the screening visit.
* LDL cholesterol >200 mg/dL as measured on the screening visit.
* Abnormal resting electrocardiogram (ECG) as measured on the screening visit: serious arrhythmias, including multifocal PVC's, frequent PVC's (defined as 10 or more per min), ventricular tachycardia (defined as runs of 3 or more successive PVC's), or sustained atrial tachyarrhythmia; 2nd or 3rd degree A-V block, QTc interval > 480 msec or other significant conduction defects.
* Presence or history of any metabolic or chronic health problems which would affect appetite, food intake, energy metabolism, or ability to participate in physical activity: cardiovascular disease (CVD), peripheral vascular disease, cerebrovascular disease, significant cardiac arrhythmias or cardiac valve disease, diabetes, uncontrolled hyper- or hypothyroidism, uncontrolled hypertension, cancer (within the last 5 years, except skin cancer or other cancers considered cured with excellent prognosis), HIV infection (unless treated with undetectable viral load), significant gastrointestinal disorders (described below), significant pulmonary disorders (described below), significant renal, musculoskeletal, neurologic, hematologic, or psychiatric disease.
* Significant gastrointestinal disorders including chronic malabsorptive conditions, active peptic ulcer disease, Crohn's disease, Ulcerative Colitis, chronic diarrhea, or active gallbladder disease.
* Significant pulmonary disorders including chronic obstructive pulmonary disease (COPD), interstitial lung disease, cystic fibrosis, or uncontrolled asthma.
* Symptoms suggestive of CVD: chest pain, shortness of breath at rest or with mild exertion, syncope.
* Primary sleep disorders including but not limited to chronic insomnia >= 3 months, untreated moderate-to-severe sleep apnea (apnea hypopnea index, AHI greater than or equal to 15), narcolepsy periodic limb movements in sleep, parasomnias including sleepwalking or night terrors, Insomnia Severity Index (ISI) Score greater than or equal to 15.

  * *Note: If we find that too many screened participants are ineligible based on AHI greater than or equal to 15, we will consider increasing AHI threshold to greater than or equal to 30 in order to improve generalizability results.
  * *Note: If we find that too many screened participants are ineligible based on ISI greater than or equal to 15, we will consider increasing ISI threshold to greater than or equal to 22 in order to improve generalizability results.

o

* Night-time shiftwork, rotating work, or other circadian disruptions and disorders (e.g., diagnosed delayed sleep-wake phase disorder).
* Regular use (greater than or equal to 2 days/wk) of prescription sleep medications (e.g., benzodiazepines, doxepin, zolpidem, trazodone, etc.).
* Regular use of other prescription or over-the-counter medications known to affect appetite, weight, sleep, or energy metabolism (e.g., lithium, stimulants, anti-psychotics, tricyclic antidepressants).
* Regular use of systemic glucocorticoids (except physiological doses for replacement therapy in adrenal insufficiency).
* Regular use of anti-obesity medications (AOMs) within the last 6 months, plans to begin AOMs in the next year.
* Previous obesity treatment with surgery or weight loss device, except: (1) liposuction and/or abdominoplasty if performed > 1 year before screening, (2) lap banding if the band has been removed > 1 year before screening, (3) intragastric balloon if the balloon has been removed > 1 year before screening (4) duodenal-jejunal bypass sleeve, if the sleeve has been removed > 1 year before screening or 5) AspireAssist or other endoscopically placed weight loss device if the device has been removed > 1 year before screening.
* Current alcohol or substance abuse.
* Nicotine use (current or quit in the past 6 months).
* History of clinically diagnosed eating disorders including anorexia nervosa, bulimia, binge eating disorder. Score >20 on the Eating Attitudes Test (EATS-26) or pattern of response on the Questionnaire of Eating and Weight Patterns (QEWP-5) suggestive of possible binge eating disorder or bulimia will require further assessment by the Study MD to determine if it is appropriate for the subject to participate in the study.
* Current severe depression or history of severe depression within the previous year, based on DSM-IV-TR criteria for Major Depressive Episode. Score > 16 on the Center for Epidemiologic Studies Depression Scale (CES-D) will require further assessment by the Study MD to determine if it is appropriate for the subject to participate in the study.
* History of other significant psychiatric illness (e.g., psychosis, schizophrenia, mania, bipolar disorder) which significantly impacts sleep or which in the opinion of the Study MD would interfere with ability to adhere to the interventions.
* Currently participating in or planning to participate in any formal weight loss programs, physical activity programs, sleep health programs, or clinical trials.
* Weight change of +/- 5 kg in past 3 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of enrollment | Baseline
  Feasibility of enrollment will be assessed by whether the study team can enroll the target sample size of n=20 individuals in the study over a 3-4 month period.
Feasibility of Outcome Measure Completion | 6 months
  Outcome measure completion will be calculated by dividing the number of participants who complete outcome measures at each timepoint by the total number enrolled.
Intervention Acceptability | 6 months
  Intervention acceptability will be assessed using validated questionnaires that assess acceptability of intervention components on a 1-5 scale.
Retention | 6 months
  Retention will be assessed by dividing the number of participants completing the 6-month study by the total number that were enrolled.

SECONDARY OUTCOMES:
Weight change (kg) | Baseline (0) - 6 Months
  Body weight will be measured using a digital scale, accurate to =/-0.1 kg, in the morning in a fasted state, at baseline, 3, and 6 months. The primary outcome will be change in weight from baseline to 6 months.
Composite sleep health score | Baseline (0) - 6 Months
  The Composite Multidimensional Sleep Health Score will be assessed at baseline, 3, and 6 months. Scores range from 0-6, with a higher score indicating better sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Catenacci, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado 80045, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Given that this research is designed to develop a novel behavioral intervention (BWL+SLEEP) and collect preliminary data to support the submission of a future grant application (by the investigative team) designed to test the weight loss efficacy of the novel intervention, only data supporting publication(s) will be made available. Subset(s) of the full, clean dataset that demonstrate the principles outlined in a resulting publication(s) will be shared in a controlled access repository. All data that can be shared will be de-identified before reaching the repository.
Time Frame: Data that can be shared will be made available at the time of associated publication(s) (data underlying peer- reviewed journal articles). Data that can be shared will be available for 3 years after the last publication.
Access Criteria: Data will be shared in a generalist repository as controlled access. Our institutional IRB currently does not allow public (open access) sharing of individual participant data. Repository access will be granted to qualified individuals within the scientific community who request access to validate and replicate the published research findings or to perform analyses that align with the research aims outlined in the approved protocol. Data users also agree not to share or redistribute any data downloads. Any publications or presentations resulting from the use of the shared dataset must appropriately acknowledge the data source, appropriately list authors (approved by Study PI), and cite the associated publications. The requester's institutional IRB or equivalent body must approve the requested use of the data. To gain access, data requestors will need to sign a data transfer agreement outlining agreement with the above conditions.